CLINICAL TRIAL: NCT06370260
Title: A Randomized Placebo-Controlled Clinical Trial Assessing the Efficacy of a Hydrogen Peroxide Gel (UNISEPT®ORAL GEL) for Oral Wound Healing, Postoperative Symptoms and Oral Hygiene in Patients Undergoing Incisional or Excisional Punch Biopsy of Gingival or Palatal Oral Mucosa
Brief Title: Assessing the Efficacy of a Hydrogen Peroxide Gel for Oral Wound Healing and Oral Hygiene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Ioulia And Irene Tseti Pharmaceutical Laboratories S.A. (Industry)
Responsible Party: Principal Investigator, Nikolaos Nikitakis, PROFESSOR AND CHAIR, DEPT. OF ORAL MEDICINE & PATHOLOGY AND HOSPITAL DENTISTRY, UNIVERSITY OF ATHENS, GREECE, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INTM-PMCF-UNIGEL; 571/13.02.2023 (Other: INTERMED S.A)
Record Dates: First submitted 2024-04-13; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Wound Heal; Postoperative Pain; Biopsy Wound; Wound; Mouth; Quality of Life; Dental Plaque; Gingival Inflammation
Keywords: oral gel; oral wound healing; oral biopsy; gingiva; palate; postoperative pain; hydrogen carbamide; hydrogen peroxide; oral hygiene; plaque index; gingival index; secondary intention healing; quality of life
MeSH Terms: conditions — Pain, Postoperative; Wounds and Injuries; Dental Plaque; Gingivitis

STUDY DESIGN:
Intervention Model Description: This trial is designed as a prospective, randomized, placebo-controlled, triple blinded, with two parallel groups and an equal allocation ratio in all groups. In this study, the intervention consists of delivery of a hydrogen carbamide/peroxide gel or placebo gel, made by the same manufacturer.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UNISEPT® ORAL GEL (Experimental): A gel containing hydrogen carbamide/peroxide as active ingredient
  Interventions: Device: Hydrogen Carbamide/Peroxide Gel
- PLACEBO (Placebo Comparator): A gel that looks and tastes like UNISEPT® ORAL GEL without active ingredients
  Interventions: Device: Placebo Gel

INTERVENTIONS:
Device: Hydrogen Carbamide/Peroxide Gel — UNISEPT® ORAL GEL is an oral gel containing 10% w/v urea peroxide which releases 3.50% w/w hydrogen peroxide, glycerin, propylene glycol, carbopol, disodium EDTA, sodium saccharin, methyl salicylate, menthol, and water, serving as the active ingredient.
  Participants should apply the gel to the biopsy area and the corresponding sextant teeth three times daily, leaving it on for five minutes without rinsing, for a total of 14 days, beginning on day 0., i.e. the day of the biopsy (see procedure in the detailed description). Consumption of liquid or solid foods should be avoided for at least thirty minutes following gel application.Participants are asked to maintain their usual oral hygiene routine.
  UNISEPT® ORAL GEL is a Class IIa, CE-marked medical device made and distributed by Intermed S.A. and Ioulia And Irene Tseti Pharmaceutical Laboratories S.A.
  Other Names: UNISEPT® ORAL GEL
  Arms: UNISEPT® ORAL GEL
Device: Placebo Gel — Placebo gel is a similar (look-and-taste-alike) product to UNISEPT® ORAL GEL, made by the same manufacturer, without active ingredients, containing glycerin, propylene glycol, carbomer, menthol, sodium saccharin, methyl salicylate, triethanolamine.
  Participants are called upon to apply the gel in exactly the same way as the experimental product, i.e apply the gel to the biopsy area and the corresponding sextant teeth three times daily, leaving it on for five minutes without rinsing, for a total of 14 days, beginning on day 0.
  Arms: PLACEBO

SUMMARY:
This study aims to assess the effectiveness and safety of a hydrogen carbamide/peroxide gel, called UNISEPT® ORAL GEL, in promoting oral wound healing, alleviating postoperative symptoms, and enhancing oral hygiene.

Study participants will include individuals with any suspicious lesion in their gums or the roof of their mouth. They will undergo a procedure to remove a small piece of tissue for testing (biopsy) in order to confirm the diagnosis.This is a standardized diagnostic procedure that involves the use of a punch, which is a plastic handpiece with a cylindrical cutting blade. Subsequently, the wound heals naturally without the need for sutures.

Researchers are comparing this gel with a placebo (a look-and-taste-alike substance that contains no active ingredients) to see if it is helpful with healing of wounds in the mouth and associated symptoms, improving oral hygiene. Participants randomly get the hydrogen carbamide/peroxide gel or the placebo one to use for 14 days after the biopsy. The researchers will not know which one they are providing as the gel tubes will be identical.

Oral wound healing, postoperative symptoms (such as pain, eating and speech difficulties), oral hygiene (dental plaque and gingival inflammation) and quality of life are assessed during a 14-day period after the biopsy. Participants are required to visit the clinic three times, one for the initial biopsy, one at 7 days and one at 14 days after the biopsy. They are asked to fill in some questionnaires, while certain procedures (taking a photo the site of the biopsy) and assessments (like evaluating the dental plaque and gingival inflammation) take place. During the first week they, also, keep a diary of their symptoms, as instructed.

DETAILED DESCRIPTION:
This is a prospective, randomized, triple-blind, placebo-controlled clinical trial and post-market clinical follow-up (PMCF) study, expected to last approximately 12 months. All procedures/visits/examinations are taking place in the Oral Medicine and Pathology Clinic at the School of Dentistry, National and Kapodistrian University of Athens, Greece. Participants, women or men, with any lesion in the gingiva or the palate (potentially malignant disorders, pigmented lesions, soft tissue masses) that require an incisional or excisional biopsy, following histopathological examination, can be enrolled, after checking if they comply with the study's criteria. Then, they are informed about the study and the biopsy procedure and they sign the Ιnformed Consent Form.

All biopsies are obtained from the gingiva or hard palate with a sterile disposable or reusable punch of 4,6 or 8mm in diameter, resulting in the extraction of similar tissue cylinders.The punch is grasped between the index and thumb, supporting the cylinder over the target lesion. Healing by secondary intention follows, as suturing of the residual wound is not necessary, and the bleeding can be contained by simply applying a piece of gauze.

Participants are instructed to have cold and soft diet for the day. Use of 500mg paracetamol up to 3 times is permitted for day 0. Following their normal oral hygiene routine (brushing and toothpaste) is suggested.

Subsequently, they are assigned randomly in a 1:1 ratio to receive either a hydrogen carbamide/peroxide gel (UNISEPT® ORAL GEL - Intermed S.A. and Ioulia And Irene Tseti Pharmaceutical Laboratories S.A) or a placebo comparator, i.e. a look-alike substance that lacks active ingredients (such as hydrogen carbamide/peroxide). Both participants and investigators are masked. Follow-up examinations are conducted at 7 and 14 days.

The evaluation includes:

oral wound healing (secondary intention) assessed by percentage healing index (PHI)(primary outcome)

and secondary outcomes: oral wound healing assessed by clinical parameters (such as redness, oidema, pus discharge) postoperative symptoms (such as pain, eating and speech difficulties) quality of life assessed by a questionnaire oral hygiene via plaque and gingival indices.

All data are anonymized and the outcome assessors are masked.

UNISEPT® ORAL GEL is a Class IIa, CE-marked (Conformité Européenne) medical device. This gel contains hydrogen carbamide that breaks down to hydrogen peroxide, which has antiseptic and antimicrobial properties. These substances have been used in wound healing either in skin or intraorally, as well as in oral hygiene for a long time. However, to date, there is no clinical trial examining the use of a hydrogen carbamide/peroxide product in oral wound healing and postoperative symptoms. Published clinical studies on the control of dental plaque and periodontal inflammation exhibit partially conflicting results.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Patients requiring incisional or excisional biopsy in the gingiva or palate
3. Patients who are legally competent and able to understand the information about the study, have been informed of the nature, scope and utility of the study, voluntarily agree to participate and have signed the consent form

Exclusion Criteria:

1. Age <18 years
2. Total number of teeth in the selected sextant <2
3. Existence of orthodontic appliances
4. Presence or history of oral malignant lesions
5. Existence of viral or other infections of the oral cavity, that could interfere with the primary outcomes of the study
6. Currently undergoing and/or has received radiation therapy to the head or neck
7. Currently receiving or has received within the previous 12 months chemotherapy and/or targeted therapies for any malignancy
8. History of acute myocardial infarction and/or vascular stroke during the last 6 months
9. Patients with poor glycemic control (HbA1c ≥ 7% within the previous 3 months according to American Diabetes Association (ADA) recommendations), uncontrolled type I or II diabetes mellitus or other systemic diseases known to affect oral wound healing
10. Use of antibiotics in the last 1 month prior to biopsy or conditions requiring antibiotic prophylaxis
11. Use of any antimicrobial mouthwash in the last 1 month before the biopsy
12. Concurrent immunocompromised status and/or use of immunosuppressant medications (e.g. corticosteroids) and steroid inhalers or nasal sprays within the last 1 month prior to enrollment
13. Malnutrition
14. Alcohol abuse and (illicit) drug use disorders
15. Pregnancy or lactation/nursing/breast feeding
16. Known allergy to any of the ingredients of the study products
17. Inability to provide informed consent
18. Participation in another study of an investigational product or device until the primary endpoint is met
19. Other medical condition that, in the opinion of the investigator, may be causing the patient's non-compliance with the clinical investigation plan or confusion in interpreting the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Assessment of wound healing based on Percentage Healing Index on day 14 | Day 14
  The Percentage Healing Index (PHI) is calculated based on three distinct values: the wound area at T0 and T2.These values are acquired through standardized pictures taken immediately after biopsy (T0) and 14 days post-biopsy (T2), with the aid of a UNC 15 (North Carolina) periodontal probe, acting as a calibrator, that was placed alongside the treated area.The images obtained are processed using software (Image J, developed by Wayne Rasband and contributors at the National Institutes of Health, USA), capable of calculating the area in square millimeters (mm).
  Initially, the T2 area is divided by the T0 area, and the result is multiplied by 100. The resulting value, known as the percentage unhealed index (PUI), indicates the percentage of the lesion that remained unhealed. The complementary value to this percentage is defined as the PHI at T2.
  Comparisons will be made between the UNISEPT® ORAL GEL versus the placebo group.
Assessment of wound healing based on Percentage Healing Index on day 7 | Day 7
  The Percentage Healing Index (PHI) is calculated based on three distinct values: the wound area at T0 and T1.These values are acquired through digital photographs taken immediately after biopsy (T0) and at 7 days post-biopsy (T1), with the aid of a periodontal probe, acting as a calibrator, that was placed alongside the treated area.The images obtained are processed using software (Image J, developed by Wayne Rasband and contributors at the National Institutes of Health, USA), capable of calculating the area in square millimeters.
  Initially, the T1 area is divided by the T0 area, and the result is multiplied by 100.The resulting value, known as the percentage unhealed index (PUI), indicates the percentage of the lesion that remained unhealed. The complementary value to this percentage is defined as the PHI at T1.
  Comparisons will be made between the UNISEPT® ORAL GEL versus the placebo group.

SECONDARY OUTCOMES:
Postoperative symptoms (pain, eating and speech difficulty) during the first week (at home) | Days 0,1,2,3,4,5 and 6
  Participants will be given a pain diary (PD) to complete at home daily at the end of the day, from day 0 to day 6, with instructions for its completion. Specifically, the participants will record: the greatest intensity of the postoperative pain, as perceived (Numerical and Visual Scale, ranked 0-10), difficulty in eating (Yes/No), difficulty in speaking (Yes/No) and whether any analgesic treatment, apart from the one recommended for day 0, has been necessary (No or Yes: Which one?). Comparisons will be made between the two groups for every day from day 0 to day 6
Postoperative symptoms (pain, eating and speech difficulty) on day 7 | Day 7
  During the visit in day 7, participants will be asked to record: the greatest intensity of the postoperative pain, as perceived (Numerical and Visual Scale, ranked 0-10), difficulty in eating (Yes/No), difficulty in speaking (Yes/No) and whether any analgesic treatment has been necessary (No or Yes: Which one?). Comparisons will be made between the two groups.
Postoperative symptoms (pain, eating and speech difficulty) on day 14 | Day 14
  During the visit in day 14, participants will be asked to record: the greatest intensity of the postoperative pain, as perceived (Numerical and Visual Scale, 0-10), difficulty in eating (Yes/No), difficulty in speaking (Yes/No) and whether any analgesic treatment has been necessary (No or Yes: Which one?). Comparisons will be made between the two groups.
Wound healing based on clinical signs | Days 7 and 14
  The researcher will record the following clinical signs after a clinical examination: redness of the biopsy area compared to the adjacent healthy tissue, presence of swelling, pus discharge, and bleeding upon palpation (Yes/No)
Oral Hygiene - Dental Plaque: Sextant Plaque Index | Days 0,7 and 14
  The Plaque Index (PI) by Silness & Loe 1964 is a score of 0-3 with higher scores indicating greater plaque accumulation. A UNC 15 periodontal probe is used. Every tooth is evaluated at 4 sites (mesiobuccal, mid-buccal, distobuccal, and lingual) as 0 = No plaque, 1 = A film of plaque adhering to free gingival margin and adjacent area of tooth, which may be seen by using the probe or disclosing solution on the tooth surface, 2 = Moderate accumulation of soft deposits within the gingival pocket, or on the tooth and gingival margin, which can be seen with the naked eye, 3 = Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  The calculation of the index refers to the sum of the measurements on the 4 surfaces of the selected sextant examined divided by four and then by the number of teeth examined. The final score ranges from 0-3. PI is measured in all visits and comparisons will be made between the two groups on day 7 and 14.
Oral Hygiene - Gingival Inflammation: Sextant Gingival Index | Days 0,7 and 14
  The Gingival Index (GI) by Loe & Silness 1963 scores from 0 to 3, with higher scores indicating greater inflammation. The examination is performed by sliding the periodontal probe (UNC 15) on the free gums (modification according to Löe - 1967) on all existing teeth of the person. Every tooth is evaluated at 4 surfaces (mesiobuccal, mid-buccal, distobuccal, and lingual). By dividing the sum of the values by 4, the gingival index of the tooth is calculated. The selected sextant gingival index is obtained by summing the indices of each tooth divided by the total number of teeth examined. The overall index score, representing inflammation, is rated as mild (mean 0,1-1,0), moderate (1,1-2,0) and severe (2,1-3). Comparisons of the GI scores will be made between the 2 groups on day 7 and 14.
Oral Health Related Quality of Life | Day 14
  The Oral Health Impact Profile-14 (OHIP-14) scale is used to measure the participants' oral health related quality of life (OHRQoL) after the procedure. It has seven conceptualized domains (two items per domain - 14 total): functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. Participants are asked to rate how frequently they experienced an oral health impact (as described by each item), scoring on a five-point Likert scale: never (score 0), hardly ever (score 1), occasionally (score 2), fairly often (score 3) and very often (score 4). Thus, OHIP-14 scores can range from 0 to 56. A high total value indicates a high negative impact on the OHRQoL. Comparisons will be made between the two groups on day 14.

OTHER OUTCOMES:
Adverse Events | Day 0,7 and 14
  Adverse events will be recorded at every visit.
Participant's comments and satisfaction regarding the provided treatment/use of the products | Day 14
  Participants are provided with a 10-item questionnaire to complete during their visit on day 14. Seven of these questions pertain to the improvement in breath odor, taste, gum health, the sensation of mouth cleanliness and freshness, as well as the reduction in gum bleeding, ease of product use, and satisfaction level resulting from product use. These are scored on a four-point Likert scale: 'not at all' (score 1), 'slightly' (score 2), 'very' (score 3), and 'extremely' (score 4). Two questions require a 'Yes' or 'No' response, inquiring whether participants would reuse the product in the event of an oral wound or ulcer and if they would recommend the product. Lastly, one question addressing compliance will be answered using a four-point Likert scale: 0-2 (score 1), 3-5 (score 2), 6-8 (score 3), and 9+ (score 4). Results will be shown for each group and comparative analyses will be conducted between the two groups.
Compliance | Day 14
  All patients are instructed to return the initially provided tube after use to record the remaining quantity. Compliance is further assessed through a question included in the aforementioned questionnaire, specifically addressing missed doses, answered on a four-point Likert scale: 0-2 (score 1), 3-5 (score 2), 6-8 (score 3), and 9+ (score 4).

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Nikitakis, DDS,MD,PHD, Study Chair — School of Dentistry, National and Kapodistrian University of Athens
Locations (1):
- Department of Oral Medicine & Pathology and Hospital Dentistry, School of Dentistry, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
The data that supports the findings of this study will be available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests will be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered.
Access Criteria: Access to trial individual participant data (IPD) can be requested by qualified investigators whose proposed research has received Institutional Review Board (IRB) approval. Data will be available via a data repository following execution of data use agreement.

REFERENCES:
- [Background] Marshall MV, Cancro LP, Fischman SL. Hydrogen peroxide: a review of its use in dentistry. J Periodontol. 1995 Sep;66(9):786-96. doi: 10.1902/jop.1995.66.9.786. PMID 7500245
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] Papagiannopoulou V, Oulis CJ, Papaioannou W, Antonogeorgos G, Yfantopoulos J. Validation of a Greek version of the oral health impact profile (OHIP-14) for use among adults. Health Qual Life Outcomes. 2012 Jan 14;10:7. doi: 10.1186/1477-7525-10-7. PMID 22244162
- [Background] Wennstrom J, Lindhe J. Effect of hydrogen peroxide on developing plaque and gingivitis in man. J Clin Periodontol. 1979 Apr;6(2):115-30. doi: 10.1111/j.1600-051x.1979.tb02190.x. PMID 379049
- [Background] Muniz FWMG, Cavagni J, Langa GPJ, Stewart B, Malheiros Z, Rosing CK. A Systematic Review of the Effect of Oral Rinsing with H2O2 on Clinical and Microbiological Parameters Related to Plaque, Gingivitis, and Microbes. Int J Dent. 2020 Oct 31;2020:8841722. doi: 10.1155/2020/8841722. eCollection 2020. PMID 33178277
- [Background] Palaia G, Tenore G, Tribolati L, Russo C, Gaimari G, Del Vecchio A, Romeo U. Evaluation of wound healing and postoperative pain after oral mucosa laser biopsy with the aid of compound with chlorhexidine and sodium hyaluronate: a randomized double blind clinical trial. Clin Oral Investig. 2019 Aug;23(8):3141-3151. doi: 10.1007/s00784-018-2735-0. Epub 2018 Oct 30. PMID 30374831
- [Background] Lopez-Jornet P, Camacho-Alonso F, Martinez-Canovas A. Clinical evaluation of polyvinylpyrrolidone sodium hyaluronate gel and 0.2% chlorhexidine gel for pain after oral mucosa biopsy: a preliminary study. J Oral Maxillofac Surg. 2010 Sep;68(9):2159-63. doi: 10.1016/j.joms.2009.09.047. Epub 2010 Jun 11. PMID 20538398